# Updated and Finalized Statistical Analysis Plan of the 'PROtective Ventilation with Higher Versus Lower PEEP During One–lung Ventilation for THORacic Surgery' (PROTHOR) Randomized Clinical Trial

The PROTHOR-investigators

#### INTRODUCTION

The 'PROtective Ventilation with High versus Low PEEP during One–lung Ventilation for THORacic surgery' (PROTHOR) randomized clinical trial compares an intraoperative ventilation strategy with higher positive end–expiratory pressure (PEEP) with recruitment maneuvers ('higher PEEP') to a conventional strategy consisting of lower PEEP of 5 cmH<sub>2</sub>O without recruitment maneuvers ('lower PEEP'), both with low tidal volumes. The primary objective of this study is to determine whether 'higher PEEP' is superior to 'lower PEEP' with regard to the incidence of postoperative pulmonary complications (PPC). Enrollment of patients in the PROTHOR study is progressing well and the study is planned to enroll the last patient in the second trimester of 2024.

To prevent outcome reporting bias and data–driven analysis results, the International Conference on Harmonization of Good Clinical Practice (ICH–GCP) recommends that clinical trials should be analyzed according to a pre–specified detailed Statistical Analysis Plan (SAP). This document presents the updated and finalized SAP of the PROTHOR study.

PROTHOR Statistical Analysis Plan (v1.0, January 17th, 2024)

#### **METHODS**

Design, ethics and registration

The PROTHOR study is an international, multicenter, parallel, two-group, prospective, randomized, patient and outcome-assessor blinded superiority clinical trial designed to determine if an intra-operative higher PEEP strategy is superior to a lower PEEP strategy with respect to the development of PPC in adult patients submitted to thoracic surgery requiring one-lung ventilation (OLV).

The protocol, with a detailed description of the study population, the two strategies and follow–up plan of the PROTHOR trial were previously published elsewhere.¹ The PROTHOR study is registered at clinicaltrials.gov (study identifier NCT02963025) and was approved by the Ethical Committee of the Istanbul University, Medical Faculty, Turkey (2016/483, April 8, 2016). Additionally, the institutional review board at the University Hospital Dresden, Technische Universität Dresden, Dresden, Germany, approved the study on 23.09.2016 (reference no. EK 392092016). The respective review boards of participating sites approved the study as well.

#### Randomization and blinding

Eligible patients are randomly allocated in a 1:1 ratio to the 'higher PEEP' or 'lower PEEP' strategy. The allocation sequence is computer—generated by an independent investigator using permuted blocks of random size of four, six, and eight patients, and stratified per center. Randomization is performed by local investigators patient—by—patient employing a dedicated, password protected, SSL—encrypted website.

At each site, at least two investigators are involved with the study. One local investigator randomizes the patients immediately before surgery, and is

responsible for the trial intervention and data collection. A second local investigator remains blinded to the assigned treatment, and is responsible for postoperative data collection.

#### **Outcomes**

The primary study outcome is a collapsed composite of PPC developing within the first five postoperative days. This endpoint follows the European Perioperative Clinical Outcome (EPCO) definition and has been used before in several clinical trials.<sup>2-4</sup> A patient that develops one or more PPCs is considered as meeting the primary outcome. The components of the composite outcome of PPC have been defined and described elsewhere,<sup>1</sup> and include: 1) aspiration pneumonitis; 2) moderate respiratory failure; 3) severe respiratory failure; 4) acute respiratory distress syndrome (ARDS); 5) pulmonary infection; 6) atelectasis; 7) cardiopulmonary edema; 8) pleural effusion; 9) pneumothorax on the non-surgical lung; 10) pulmonary infiltrates; 11) prolonged air leakage; 12) purulent pleuritic; 13) pulmonary embolism; and 14) lung hemorrhage. The selected PPC can sensibly be merged as they share common pathophysiological mechanisms and have plausibility to be affected in the same direction by the intervention tested in this study.

Secondary outcomes include: 1) extended PPC, including bronchospasm or mild respiratory failure; 2) severe PPC, as defined in a recent published clinical trial<sup>5</sup> (composite of severe respiratory failure, pneumothorax, ARDS, pulmonary infection, prolonged air leakage, purulent pleuritis, new requirement of non-invasive or invasive ventilation due to respiratory failure and/or atelectasis); 3) a composite outcome of intraoperative complications, including use of continuous positive airway pressure for the non-ventilated lung, use of inhaled nitric

oxide/prostacycline, use of selective fiberoscope insufflation, hypotension unresponsive to fluids and/or vasoactive drugs, new arrhythmias unresponsive to intervention, need for high dosage of vasoactive drugs, need for massive transfusion, life-threatening surgical complication (including major bleeding, tension pneumothorax and intracranial injury), hypoxemia and hypercapnia rescue maneuvers; 4) postoperative extrapulmonary complications, including systemic inflammatory response syndrome, sepsis, severe sepsis, septic shock, extrapulmonary infection, coma, acute myocardial infarction, acute renal failure. disseminated intravascular coagulation, stroke, hepatic failure, and gastrointestinal failure; 5) need for unexpected intensive care unit admission or readmission; 6) any postoperative respiratory intervention used for respiratory failure (new requirement of non-invasive ventilation or mechanical ventilation); 7) number of hospital-free days at day 28; 8) in-hospital mortality; 9) 90-day mortality; 10) arterial blood gas analysis during surgery (PaO<sub>2</sub>, PaCO<sub>2</sub>, pHa). All definitions are available in Table 1.

#### Cleaning and closing of the database

The database will be locked as soon as all data are entered and all discrepant or missing data are resolved, after all efforts are employed to fix missing data, complete the database, and we consider that the remaining issues cannot be fixed. At this step, the data will be reviewed before database locking. After locking, the data will be exported for statistical analysis. At this stage, permission for access to the database will be removed for all investigators, and the database is archived.

#### Missing data

No or minimal losses to follow–up for the primary outcome is anticipated. Complete–case analysis will be carried out for all outcomes. However, if more than 5% of missing data is found for the primary outcome, a sensitivity analysis using multiple imputations and estimating–equation methods will be carried out. Multiple imputation will consider imputation models based on prognostic baseline and post–baseline variables under a missing at random assumption.

#### Sample size

An adaptive trial design is used, which accumulates data and uses external information to modify aspects of the design without undermining the validity and integrity of the trial. The group sequential methods design offers the possibility for early stopping the study if the experimental treatment shows a statistically significant therapeutic advantage at an interim assessment, but also allows early stopping for futility if the interim analysis reveals that, with high probability, the trial will be negative.

PROTHOR is designed to enroll a total of 2378 patients (1189 in each arm). This number allows the detection of a reduction in the incidence of the primary outcome from 23% in the 'lower PEEP' group to 17.25% in the 'higher PEEP' group (relative risk reduction of 25%), considering a type I error of 5%, a power of 90%, similar allocation ratio between the arms (1:1) and a dropout rate of 5%. The required sample size is calculated based on an estimated effect size derived from individual patient data from previous trials, <sup>3,4,6-9</sup> and the LAS VEGAS study. <sup>10</sup>

An alpha–spending function was used to generate efficacy boundaries and a beta-spending function to generate futility boundaries (gamma family spending function, type I error 0.05, type II error 0.1). By using a gamma of -4 for the alpha

and gamma of -2 for the beta spending function a moderate hurdle for early stopping for efficacy and a reasonable chance to stop early due to futility is considered. A non-binding futility boundary was constructed in such a way that it can be overruled if desired without inflating the type 1 error. This flexibility is important, since the data monitoring committee might well prefer to keep the trial going to gather additional information, despite crossing the futility boundary (**Figure 1** and **Table 2**).

#### Interim analyses

Five interim assessments for evaluation of efficacy, harm, and/or futility were planned, with the aim of possibly stopping the study early. The planned number of assessments describes the number of time points, including the closing date of the study, at which the investigator plans to analyze the thus far collected data. The spacing of assessments will be equal. Therefore, interim analyses were performed after 20% (476 patients), 40% (952 patients), 60% (1426 patients), and 80% (1902 patients) of the planned inclusions, and the final analysis will be performed after 2378 patients (100%) are included (**Table 2**).

#### Statistical analyses

All statistical analyses will be conducted on an intention—to—treat basis, with patients analyzed according to their assigned treatment arms, except for cases lost to follow up or withdrawal of informed consent. In addition, a per—protocol analysis will be conducted. Variables will be expressed as counts and percentages, means and standard deviations (SD), or medians and interquartile ranges (IQR) whenever appropriate.

The study was designed to detect a difference in the primary outcome with 90% power, using a two–sided superiority hypothesis test with a significance level

of 0.0428 (correspondent to the Z-value of 2.025 for efficacy or futility in the final analysis in **Table 2**) and presented with a two–sided 95% confidence interval. Secondary outcomes will be assessed using a two–sided superiority hypothesis test with a significance level of 0.05 and presented with a two–sided 95% confidence interval. In addition to the unadjusted *p* values for secondary outcomes, a Holm–Bonferroni procedure will be applied to control for multiple testing. Analyses will be performed using the software R (R Core Team, 2016, Vienna, Austria). A list of proposed tables and figures is in **Table 3**.

#### Trial profile

Patient flows will be represented in a CONSORT flowchart (Proposed Inserts).

#### Baseline characteristics

A description of the baseline characteristics of the trial participants will be presented by treatment group (**Proposed Inserts**). Discrete variables will be summarized as numbers (%). Percentages will be calculated according to the number of trial participants for whom data are available. Whenever values are missing, the denominator will be stated in the table and no assumptions or imputations will be made. Continuous variables will be summarized by either mean and standard deviation (SD) or median and interquartile range (IQR), according to the observed distribution of the variable.

#### Adherence to study protocol and ventilatory variables

Surgical and perioperative characteristics will be reported (**Proposed Inserts**). Ventilatory variables and vital signs will be reported after intubation, one hour, and in the last hour of surgery and compared between the two groups. Absolute differences between groups will be calculated using median regression for continuous variables (reported as median difference) and generalized linear

models with binomial distribution and an identity link for binary variables (reported as difference in percentages). Plots comparing ventilatory variables and vital signs among the groups during the first three hours of surgery and in the last hour will be drawn (presenting the data as mean and 95% confidence interval in each time point).

#### Other daily characteristics

Daily variables will be reported according to the description in **Proposed Inserts**. Absolute differences between groups will be calculated using median regression for continuous variables (reported as median difference) and generalized linear models with binomial distribution and an identity link for binary variables (reported as difference in percentages). Plots comparing daily variables among the groups will be constructed (presenting the data as mean and 95% confidence interval in each time point).

#### Primary outcome

The effect of 'higher PEEP' compared to 'lower PEEP' on the incidence of PPC will be assessed using a mixed–effect generalized linear model with binomial distribution and identity link, with sites included as random effects to account for the clustering effect and reported as absolute difference with a two–sided 95% confidence interval. Results will be presented in a table of outcomes (**Proposed Inserts**).

#### Secondary outcomes

For binary outcomes, the effect of 'higher PEEP' compared to 'lower PEEP' will be assessed using a mixed-effect generalized linear model with binomial distribution and identity link, with sites included as random effects to account for the clustering effect and reported as absolute difference with a two-sided 95%

confidence interval. For continuous outcomes, the comparison will be made using a mixed-effect median regression with sites also including as clustering effect, and reported as median difference with a two–sided 95% confidence interval. 90-day mortality will be assessed using Kaplan–Meier curves, and hazard ratios with 95% confidence intervals will be calculated with (shared-frailty) Cox proportional hazard models without adjustment for covariates and including sites as frailty. The proportional hazard assumptions will be tested using scaled Schoenfeld residuals and alternative parametric survival models will be used if the proportionality assumption is not sustained. In addition, a Holm–Bonferroni correction to control the family–wide error rate to the *p* values for all secondary outcomes will be done and presented in a Table.

#### Per-protocol analysis

The per–protocol population will consist of patients truly ventilated according to the protocol. Thus, patients will be excluded from this population if receiving PEEP < 10 cm  $H_2O$  in the 'higher PEEP' group or PEEP > 5 cm  $H_2O$  and  $FiO_2$  < 1.0 in the 'lower PEEP' group, unless rescue for hypoxemia or hypercapnia required adjustments of PEEP and  $F_iO_2$  as defined by the protocol.

#### Subgroup analysis

Treatment effects on incidence of PPC will be analyzed according to the following predefined subgroups: 1) type of surgery (non–thoracoscopic versus thoracoscopic); 2) positioning (lateral decubitus versus supine position); 3) baseline  $SpO_2 < 96\%$  versus  $SpO_2 \ge 96\%$ ; 4) chronic obstructive pulmonary disease (COPD) versus non-COPD; 5) body mass index < 30 kg/m² versus  $\ge$  30 kg/m²; and 6) duration of one-lung ventilation < 120 versus  $\ge$  120 minutes. Analyses of heterogeneity of effects across subgroups will be performed with the

use of treatment-by-subgroup term added to the primary model and will be presented in a forest plot.

#### Other exploratory analyses

Given that the primary outcome of the present study is a collapsed composite, the choice of the statistical method is an important part of designing since various methods provide different power, depending on the situation. In addition to the standard analysis described above, the following analyses will be performed:

- Count analysis: the number of positive component events (i.e., 'count')
  across the composite will be assessed. The groups will be compared on
  the count using a Wilcoxon rank sum test, and the odds ratio with the 95%
  confidence interval will be assessed with a cumulative logistic regression
  model;
- Individual component analysis: the effect of the intervention in each component will be analyzed estimating the risk ratio and confidence intervals with Wald's likelihood ratio approximation test using a Bonferroni correction for multiple comparisons. The 99.6% Bonferroni—corrected confidence intervals will be reported (1 0.05/14 = 0.996);
- Common effect test: A multivariate (i.e., multiple outcomes per subject)
   generalized estimating equations (GEE) model will be used to estimate a
   common effect odds ratio across the components;
- Average relative effect test: The average relative effect test will be
  assessed by averaging the component-specific treatment effect from the
  distinct effects model, and testing whether the average is equal to zero. In
  the GEE distinct effect model a distinct treatment effect is estimated for
  each component; and

PROTHOR Statistical Analysis Plan (v1.0, January 17th, 2024)

 Heterogeneity of treatment effect: Heterogeneity of treatment effect across components will be assessed by a treatment-by-component interaction test in the distinct effects GEE model.

#### **REFERENCES**

- 1. Kiss T, Wittenstein J, Becker C, et al. Protective ventilation with high versus low positive end-expiratory pressure during one-lung ventilation for thoracic surgery (PROTHOR): study protocol for a randomized controlled trial. Trials 2019;20:213.
- 2. Jammer I, Wickboldt N, Sander M, et al. Standards for definitions and use of outcome measures for clinical effectiveness research in perioperative medicine: European Perioperative Clinical Outcome (EPCO) definitions: a statement from the ESA-ESICM joint taskforce on perioperative outcome measures. Eur J Anaesthesiol 2015;32:88–105.
- 3. Hemmes SN, Gama de Abreu M, Pelosi P, Schultz M. High versus low positive end-expiratory pressure during general anaesthesia for open abdominal surgery (PROVHILO trial): a multicentre randomised controlled trial. Lancet 2014;384:495–503.
- 4. Ferrando C, Soro M, Unzueta C, et al. Individualised perioperative openlung approach versus standard protective ventilation in abdominal surgery (iPROVE): a randomised controlled trial. Lancet Respir Med 2018;6:193–203.
- 5. Ferrando C, Carramiñana A, Piñeiro P, et al. Individualised, perioperative open-lung ventilation strategy during one-lung ventilation (iPROVE-OLV): a multicentre, randomised, controlled clinical trial. Lancet Respir Med 2023;[in press].
- 6. Futier E, Constantin JM, Paugam-Burtz C, et al. A trial of intraoperative low-tidal-volume ventilation in abdominal surgery. N Engl J Med 2013;369:428–37.

- 7. Ge Y, Yuan L, Jiang X, Wang X, Xu R, Ma W. Effect of lung protection mechanical ventilation on respiratory function in the elderly undergoing spinal fusion. J Cent South Univ 2013;38:81–5.
- 8. Severgnini P, Selmo G, Lanza C, et al. Protective mechanical ventilation during general anesthesia for open abdominal surgery improves postoperative pulmonary function. Anesthesiology 2013;118:1307–21.
- 9. Ferrando C, Soro M, Unzueta C, et al. Rationale and study design for an individualised perioperative open-lung ventilatory strategy with a high versus conventional inspiratory oxygen fraction (iPROVE-O2) and its effects on surgical site infection: study protocol for a randomised controlled trial. BMJ Open 2017;7:e016765.
- 10. LAS VEGAS Investigators. Epidemiology, practice of ventilation and outcome for patients at increased risk of postoperative pulmonary complications: LAS VEGAS an observational study in 29 countries. Eur J Anaesthesiol 2017; 34:492–507.
- 11. Holm S. A simple sequentially rejective multiple test procedure. Scand J Stat 1979; 6:65-70.

Table 1 - Definitions of Outcomes

| Outcomes | Definition |
|---|---|
| Aspiration pneumonitis | Respiratory failure after the inhalation of regurgitated gastric contents. |
| Moderate respiratory failure | $SpO_2 < 90\%$ or $PaO_2 < 60$ mmHg for 10 min in room air, responding to oxygen > 2 L/min. |
| Severe respiratory failure | Need for noninvasive or invasive mechanical ventilation due to poor oxygenation. |
| Acute respiratory distress syndrome | According to the Berlin criteria for acute respiratory distress syndrome*. |
| Pulmonary infection | Defined as new or progressive radiographic infiltrate plus at least two of the following: • Antibiotic treatment; • Tympanic temperature > 38 °C; • Leukocytosis or leucopenia (white blood cell count < 4000 cells/mm3 or > 12,000 cells/mm3); • Purulent secretions |
| Atelectasis | Lung opacification with shift of the mediastinum, hilum, or<br>hemidiaphragm towards the affected area, and<br>compensatory overinflation in the adjacent non-<br>atelectatic lung. |
| Cardiopulmonary edema | Clinical signs of congestion, including dyspnea, edema, rales and jugular venous distention, with the chest radiograph demonstrating increase in vascular markings and diffuse alveolar interstitial infiltrates. |
| Pleural effusion | Chest x-ray demonstrating blunting of the costophrenic angle, loss of the sharp silhouette of the ipsilateral hemidiaphragm in upright position, evidence of displacement of adjacent anatomical structures, or (in supine position) a hazy opacity in one hemithorax with preserved vascular shadows. |
| Pneumothorax | Air in the pleural space with no vascular bed surrounding the visceral pleura on chest radiography. |
| Pulmonary infiltrates | Chest x-ray demonstrating new unilateral or bilateral infiltrate without other clinical signs. |
| Prolonged air leakage | Air leak requiring at least 7 days of postoperative chest tube drainage. |
| Purulent pleuritic | Receiving antibiotics for a suspected infection, as far as not explained by the preoperative patient condition alone. |
| Pulmonary embolism | As documented by pulmonary arteriogram or autopsy, or supported by ventilation/perfusion radioisotope scans, or documented by echocardiography and receiving specific therapy. |
| Lung hemorrhage | Bleeding through the chest tubes requiring reoperation, or three or more red blood cell packs. |
| Bronchospasm | Newly detected expiratory wheezing treated with bronchodilators. |
| Mild respiratory failure | $PaO_2 < 60$ mmHg (or < 7.9 kPa) or $SpO_2 < 90\%$ for 10 minutes in room air, but responding to oxygen $\leq 2$ L/min. |
| Systemic inflammatory response syndrome | <ul> <li>Presence of two or more of the following:</li> <li>Body temperature &lt; 36 °C or &gt; 38 °C;</li> <li>Heart rate &gt; 90 beats per minute;</li> <li>Respiratory rate &gt; 20 breaths per minute or, on blood gas, a PaCO<sub>2</sub> &lt; 32 mmHg (4.3 kPa);</li> <li>White blood cell count &lt; 4000 cells/mm3 or &gt; 12,000 cells/mm3, or &gt; 10% band forms.</li> </ul> |
| Sepsis | Systemic inflammatory response syndrome in response to a confirmed infectious process; infection can be suspected or proven (by culture, stain, or polymerase |

| | chain reaction), or a clinical syndrome pathognomonic for infection |
|---|---|
| Severe sepsis | Sepsis with organ dysfunction, hypoperfusion, or hypotension), septic shock (sepsis with refractory arterial hypotension or hypoperfusion abnormalities in spite of adequate fluid resuscitation); signs of systemic hypoperfusion may be either end-organ dysfunction or serum lactate greater than 4 mmol/dL, other signs include oliguria and altered mental status. |
| Septic shock | Sepsis plus hypotension after aggressive fluid resuscitation, typically upwards of 6 L or 40 mL/kg of crystalloid. |
| Extrapulmonary infection | Wound infection + any other infection. |
| Coma | Glasgow Coma Score < 8 in the absence of therapeutic coma or sedation. |
| Acute myocardial infarction | Detection of rise and/or fall of cardiac markers (preferably troponin) with at least one value above the 99th percentile of the upper reference limit, together with symptoms of ischemia, electrocardiography changes indicative of new ischemia, development of pathological Q-waves, or imaging evidence of new loss of viable myocardium or new regional wall motion abnormality or sudden unexpected cardiac death, involving cardiac arrest with symptoms suggestive of cardiac ischemia (but death occurring before the appearance of cardiac markers in blood). |
| Acute renal failure | <ul> <li>Risk: increased creatinine × 1.5 or glomerular filtration rate (GFR) decrease &gt; 25% or urine output (UO) &lt; 0.5 mL/kg/h × 6 h;</li> <li>Injury: increased creatinine × 2 or GFR decrease &gt; 50% or UO &lt; 0.5 mL/kg/h × 12 h;</li> <li>Failure: increased creatinine × 3 or GFR decrease &gt; 75% or UO &lt; 0.3 mL/kg/h × 24 h or anuria × 12 h;</li> <li>Loss: persistent acute renal failure = complete loss of kidney function &gt; 4 weeks.</li> </ul> |
| Disseminated intravascular coagulation | <ul> <li>Platelet count &lt; 50 (2 points), &lt; 100 (1 point), or ≥ 100 (0 points);</li> <li>D-dimer &gt; 4 μg/mL (2 points), &gt; 0.39 μg/mL (1 point) or ≤ 0.39 μg/mL (0 points);</li> <li>Prothrombin time &gt; 20.5 s (2 points), &gt; 17.5 s (1 point), or ≤ 17.5 s (0 points).</li> <li>If ≥ 5 points: overt disseminated intravascular coagulation</li> </ul> |
| Stroke | New clinical signs of stroke lasting longer than 24 h and corresponding findings in radiologic imaging |
| Hepatic failure | Hepatic failure during short-term follow-up (5 postoperative days) is considered as follows: • Bilirubin serum level > 2 mg/dL; • Elevation of alanine amino transferase/aspartate amino transferase; • Lactate dehydrogenase × 2 above normal values. During long-term follow-up (until postoperative day 90): • New presence of hepatic encephalopathy; • Coagulopathy (international normalized ratio (INR) > 1.5) within 8 weeks after initial signs of liver injury (e.g., jaundice) without evidence for chronic liver disease. |

#### PROTHOR Statistical Analysis Plan (v1.0, January 17th, 2024)

| | Any type of gastrointestinal bleeding or gastrointestinal failure score documented as follows: |
|---|---|
| | <ul> <li>0 = normal gastrointestinal function;</li> </ul> |
| | <ul> <li>1 = enteral feeding with under 50% of calculated</li> </ul> |
| | needs or no feeding 3 days after abdominal |
| Gastrointestinal failure | surgery; |
| | <ul> <li>2 = food intolerance or intraabdominal</li> </ul> |
| | hypertension; |
| | • 3 = food intolerance and intra-abdominal |
| | hypertension; and |
| | <ul> <li>4 = abdominal compartment syndrome</li> </ul> |
| | Defined as the number of days that a patient was not in |
| | hospital nor rehabilitation or nursing facility at day 28 after |
| | randomization. Hospital readmission is only counted if the |
| Number of hospital-free days at day 28 | patient stays overnight (= 2 days). Patients who die or |
| | have longer length of stay than 28 days are assigned zero |

<sup>\*</sup> ARDS Definition Task Force, Ranieri VM, Rubenfeld GD, et al. Acute respiratory distress syndrome: the Berlin Definition. JAMA 2012;307:2526-33.

hospital free days.

Table 2 – Z-statistic Boundaries and Boundary Crossing Probabilities

| I OOK | Information<br>Fraction | Ν | Cumulative | Z-efficacy/harm | Z-futility | Boundary crossing<br>probabilities under H₁ | | |
|---|---|---|---|---|---|---|---|---|
| | Fraction | | α spent | β spent | - | _ | Efficacy | Futility |
| 1 | 0.20 | 452 | 0.001 | 0.008 | ± 3.252 | ± 0.031 | 0.042 | 0.008 |
| 2 | 0.40 | 904 | 0.004 | 0.019 | ± 2.986 | ± 0.152 | 0.170 | 0.011 |
| 3 | 0.60 | 1355 | 0.009 | 0.036 | ± 2.692 | ± 0.631 | 0.281 | 0.017 |
| 4 | 0.80 | 1807 | 0.022 | 0.062 | ± 2.374 | ± 1.344 | 0.263 | 0.026 |
| 5 | 1.00 | 2259 | 0.050 | 0.100 | ± 2.025 | ± 2.025 | 0.143 | 0.038 |

Values were calculated using power = 0.90, alpha = 0.05, gamma spending function - 4 for the alpha and - 2 for the beta, expected incidence of postoperative pulmonary complications of 23% and 17.25% in the lower and higher positive end-expiratory pressure groups, respectively. Number of patients (N) is shown without correcting for dropouts. Look, interim analysis; H1, hypothesis 1 (group difference exists).

Table 3 - List of proposed tables and figures

| | Description |
|---|---|
| Main paper | <u> </u> |
| Table 1 | Baseline Characteristics of the Included Patients |
| Table 2 | Ventilation and Intraoperative Characteristics |
| Table 3 | Primary and Secondary Outcomes |
| Figure 1 | Participant Flow Diagram |
| Figure 2 | Postoperative Pulmonary Complications in Prespecified Subgroups A forest plot showing the absolute difference and two–sided 95% confidence intervals with p value for interaction calculated via a test for treatment–by–subgroup interaction in the regression model. A solid line of reference in the number 1 and a dashed line of reference in the overall effect will be shown. |
| Online Supp | ement |
| eTable 1 | Rate of Missing Data A table showing the rate of missing data. |
| eTable 2 | Additional Baseline Characteristics A table showing additional baseline characteristics. |
| eTable 3 | Additional Intraoperative Characteristics A table showing additional intraoperative characteristics. |
| eTable 4 | Intraoperative Fluid and Drug Therapy A table reporting intraoperative fluid and drug therapy each arm. |
| eTable 5 | Protocol Deviations A table describing protocol deviations. |
| eTable 6 | Daily Assessment of Included Patients A table describing daily assessment of patients. |
| eTable 7 | Additional Daily Assessment of Included Patients A table describing daily assessment of patients. |
| eTable 8 | Daily Signs and Laboratory of Included Patients A table describing daily assessment of patients. |
| eTable 9 | Day 1 Fluid and Drug Therapy A table reporting day 1 fluid and drug therapy each arm. |
| eTable 10 | Multiplicity adjustment for secondary outcome analyses A table showing the observed p values for all the secondary outcomes and ordered from the lower until the higher and the corrected p values using a Holm–Bonferroni correction |
| eTable 11 | Sensitivity Analyses for the Primary Outcome A table showing the proposed sensitivity analyses for the primary outcome (count analysis, common effect test, average relative effect test and heterogeneity of treatment effect) |
| eFigure 1 | Tidal Volume, PEEP, Peak Pressure, Plateau Pressure, Driving Pressure and FiO <sub>2</sub> During Surgery Line graph reporting the mean and 95% confidence interval of the variables at induction, final positioning with two lung ventilation, 10 minutes of one lung ventilation and at the end of surgery by treatment group. |
| eFigure 2 | VAS Dyspnea, VAS Thoracic Pain, VAS Coughing Pain, Respiratory Rate, SpO <sub>2</sub> and Mean Arterial Pressure During the First Five Days of Follow-Up Line graph reporting the mean and 95% confidence interval of the variables in the first five days of follow-up by treatment group. |

#### PROTHOR Statistical Analysis Plan (v1.0, January 17th, 2024)

| eFigure 3 | Results of the Sensitivity Analyses for the Primary Outcome Forest plot reporting the results of all sensitivity analyses |
|---|---|
|---|---|

Futility

Efficacy

Number of included patients

Figure 1 – PROTHOR Adaptive Design

Effect size (Z) according to enrollment of patients in the PROTHOR trial (including dropouts). Values of Z were from an adaptive sequential design (see text) with stopping criteria for harm, futility, and efficacy of the intervention.

### MODIFICATIONS FROM THE ORIGINAL ANALYSIS PLAN

| ANALYSIS | ORIGINAL PLAN<br>( <i>TRIALS</i> 2019; 20:213) | UPDATE IN THE SAP*<br>(Closed in January 17 <sup>th</sup> , 2024) |
|---|---|---|
| Definition of intraoperative complications (secondary outcome) | Included 'deviation from prescribed PEEP or tidal volume' in the definition | 'deviation from prescribed PEEP or tidal volume' removed from the definition |
| Requirement of postoperative respiratory intervention (secondary outcome) | Any requirement of postoperative respiratory intervention | Requirement of postoperative respiratory intervention for respiratory failure only (excludes for reoperation) |
| Secondary outcome | | Addition of severe postoperative pulmonary complications. |
| Model for the primary outcome | Risk ratio and 95% confidence intervals calculated with Wald's likelihood ratio approximation test and with $\chi^2$ tests for hypothesis testing. | Mixed-effect generalized linear model with binomial distribution and identity link, with sites included as random effects to account for the clustering effect and reported as absolute difference with a two-sided 95% confidence interval. |
| Model for binary secondary outcomes | Risk ratio and 95% confidence intervals calculated with Wald's likelihood ratio approximation test and with $\chi^2$ tests for hypothesis testing. | Mixed-effect generalized linear model with binomial distribution and identity link, with sites included as random effects to account for the clustering effect and reported as absolute difference with a two-sided 95% confidence interval. |
| Model for hospital-free<br>days at day 28 | Student <i>t</i> test and reported as the mean difference between the two groups. The consistency of the findings of the Student <i>t</i> test will be confirmed according to the mean ratio calculated by a generalized additive model considering a zero-inflated beta distribution. | Mixed-effect median regression with sites also including as clustering effect, and reported as median difference with a two-sided 95% confidence interval. |
| Time-to-event analyses<br>for PPC | Kaplan–Meier curves will be used to report time to postoperative pulmonary complications, and hazard ratios with a 95% confidence interval will be calculated with Cox proportional hazard models without adjustment for covariates. | No time-to-event analysis planned to be performed for PPC. |
| Time-to-event analyses for 90-day mortality | Hazard ratios with 95% confidence intervals will be calculated with Cox proportional hazard models without adjustment for covariates and including sites as frailty. | Hazard ratios with 95% confidence intervals will be calculated with (shared-frailty) Cox proportional hazard models without adjustment for covariates and including sites as frailty. |
| Subgroup analysis (definition) | | Added two additional subgroups: body mass index and duration of one-lung ventilation. |
| Subgroup analysis<br>(method) | The effects on subgroups will be evaluated according to the interaction effects between each subgroup and the study arms by generalized linear models and presented in a forest plot. | Analyses of heterogeneity of effects across subgroups will be performed with the use of treatment-by-subgroup term added to the primary model and will be presented in a forest plot. |

## LIST OF PROPOSED INSERTS

Table 1 - Baseline Characteristics of the Included Patients

| Table 1 – Baseline Characteristics ( | | |
|-----------------------------------------|-------------|------------|
| | Higher PEEP | Lower PEEP |
| _ | (n = ) | (n = ) |
| Age, years | | |
| Age ≥ 65 years – no. (%) | | |
| Female gender – no. (%) | | |
| Body mass index, kg/m <sup>2</sup> | | |
| Body mass index ≥ 30 kg/m² | | |
| ARISCAT score | | |
| ARISCAT ≥ 45 – no. (%) | | |
| ASA physical status- no. (%) | | |
| 1 | | |
| 2 | | |
| 3 | | |
| 4 | | |
| Priority of surgery – no. (%) | | |
| Elective | | |
| Urgent | | |
| Emergency | | |
| Surgical procedure – no. (%) | | |
| Thoracoscopic | | |
| Open | | |
| Converted from thoracoscopic to open | | |
| Cumulated ambulation score | | |
| Co-existing disorders – no. (%) | | |
| Hypertension | | |
| Heart failure | | |
| Coronary artery disease | | |
| Diabetes | | |
| Obstructive sleep apnea | | |
| Chronic obstructive pulmonary disease | | |
| Use of noninvasive ventilation | | |
| Active cancer | | |
| Respiratory infection within last month | | |
| Smoking status | | |
| Never | | |
| Former (cessation > 3 months) | | |
| Current | | |
| Alcohol (> 2 drinks/day) | | |
| Preoperative signs | | |
| SpO <sub>2</sub> , % | | |
| Respiratory rate, breaths/min | | |
| Heart rate, beats per minute | | |
| Mean arterial blood pressure, mmHg | | |

Data are median (quartile 25th - quartile 75th) or N / total (%).
Abbreviations: PEEP is positive end-expiratory pressure; ARISCAT is The Assess Respiratory Risk in Surgical Patients in Catalonia; ASA is American Society of Anesthesiology; SpO2 is pulse oximetry.

p value

| | Higher PEEP | Lower PEEP | Absolute Difference |
|---|---|---|---|
| _ | (n = ) | (n = ) | (95% CI) |
| Recruitment maneuver – no. (%) | | | |
| Number of recruitment maneuvers | | | |
| Tidal volume, mL/kg PBW | | | |
| Induction | | | |
| Final position with two lung ventilation | | | |
| 10 minutes after one lung ventilation | | | |
| End of surgery, supine, two lung ventilation | | | |
| PEEP, cmH <sub>2</sub> O | | | |
| Induction | | | |
| Final position with two lung ventilation | | | |
| 10 minutes after one lung ventilation | | | |
| End of surgery, supine, two lung ventilation | | | |
| Peak pressure, cmH <sub>2</sub> O | | | |
| Induction | | | |
| Final position with two lung ventilation | | | |
| 10 minutes after one lung ventilation | | | |
| End of surgery, supine, two lung ventilation | | | |
| Plateau pressure, cmH₂O | | | |
| Induction | | | |
| Final position with two lung ventilation | | | |
| 10 minutes after one lung ventilation | | | |
| End of surgery, supine, two lung ventilation | | | |
| Driving pressure, cmH <sub>2</sub> O | | | |
| Induction | | | |
| Final position with two lung ventilation | | | |
| 10 minutes after one lung ventilation | | | |
| End of surgery, supine, two lung ventilation | | | |
| Respiratory rate, breaths/min | | | |
| Induction | | | |
| Final position with two lung ventilation | | | |
| 10 minutes after one lung ventilation | | | |
| End of surgery, supine, two lung ventilation | | | |
| FiO <sub>2</sub> | | | |
| Induction | | | |
| Final position with two lung ventilation | | | |
| 10 minutes after one lung ventilation | | | |
| End of surgery, supine, two lung ventilation | | | |
| SpO <sub>2</sub> , % | | | |
| Induction | | | |
| Final position with two lung ventilation | | | |
| 10 minutes after one lung ventilation | | | |
| Final of assessment assessment for a large state of the second | | | |

End of surgery, supine, two lung ventilation

Table 2 - Ventilation and Intraoperative Characteristics

| | Higher PEEP<br>(n = ) | Lower PEEP<br>(n = ) | Absolute Difference<br>(95% CI) | p value |
|---|---|---|---|---|
| etCO <sub>2</sub> , mmHg | | | | |
| Induction | | | | |
| Final position with two lung ventilation | | | | |
| 10 minutes after one lung ventilation | | | | |
| End of surgery, supine, two lung ventilation | | | | |
| Mean arterial pressure, mmHg | | | | |
| Induction | | | | |
| Final position with two lung ventilation | | | | |
| 10 minutes after one lung ventilation | | | | |
| End of surgery, supine, two lung ventilation | | | | |
| Duration of anesthesia, min | | | | |
| Duration of one lung ventilation, min | | | | |
| Duration of two lung ventilation, min | | | | |
| Duration of surgery, min | | | | |
| Duration of surgery ≥ 180 min – no. (%) | | | | |
| Fluids | | | | |
| Total intake, mL | | | | |
| Fluid balance, mL | | | | |

Data are median (quartile 25th - quartile 75th) or N / total (%).

Abbreviation: PEEP is positive end-expiratory pressure; PBW is predicted body weight;  $FiO_2$  is inspired fraction of oxygen;  $SpO_2$  is pulse oximetry;  $etCO_2$  is end-tidal carbon dioxide.

**Table 3 – Primary and Secondary outcomes** 

| Higher PEEP | Lower PEEP | Absolute Difference | n volue |
|-------------|------------|---------------------|----------------|
| (n = ) | (n = ) | (95% CI) | <i>p</i> value |

#### **Primary outcome**

Postoperative pulmonary complications – no. (%)

Aspiration pneumonitis

Moderate respiratory failure

Severe respiratory failure

Acute respiratory distress syndrome

Pulmonary infection

Atelectasis

Cardiopulmonary edema

Pleural effusion

Pneumothorax

Pulmonary infiltrates

Prolonged air leakage

Purulent pleuritic

Pulmonary embolism

Lung hemorrhage

#### **Secondary outcomes**

Extended postoperative pulmonary complications – no. (%)

Mild respiratory failure

Bronchospasm

Intraoperative complications – no. (%)

CPAP for the non-ventilated lung

iNO, prostacycline or selective fiberoscope insufflation

Hypotension unresponsive to fluids or vasoactive drugs

New arrhythmias unresponsive to intervention

#### PROTHOR Statistical Analysis Plan (v1.0, January 17th, 2024)

Need for high dosage of vasoactive drugs

Need for massive transfusion

Life-threatening surgical complication\*

Hypoxemia rescue maneuvers

Hypercapnia rescue maneuvers

Postoperative extrapulmonary complications – no. (%)

Systemic inflammatory response syndrome

Sepsis

Severe sepsis

Septic shock

Extrapulmonary infection

Coma

Acute myocardial infarction

Acute renal failure

Disseminated intravascular coagulation

Stroke

Hepatic failure

Gastrointestinal failure

Unexpected ICU admission or readmission - no. (%)

Postoperative respiratory intervention – no. (%)

Non-invasive ventilation

Invasive ventilation

Number of hospital-free days at day 28

All-cause hospital mortality – no. (%)

90-day mortality – no. (%)

Data are median (quartile 25th - quartile 75th) or N / total (%).

Abbreviations: PEEP is positive end-expiratory pressure; CPAP is continuous positive airway pressure; iNO is inhaled nitric oxide; ICU is intensive care unit.

<sup>\*</sup> Including major bleeding, tension pneumothorax and intracranial injury.

#### eTable 2 – Additional Baseline Characteristics

| e lable 2 – Additional Baseline Characteristics | | |
|---|---|---|
| | Higher PEEP | Lower PEEP |
| | (n = ) | (n = ) |
| Cumulated ambulation score | | |
| Transfer from supine-to-sitting-to-supine – no. (%) | | |
| Unable to perform function despite assistance from 2 people | | |
| Only able to perform function with assistance from 1 or 2 people | | |
| Able to perform function independently | | |
| Transfer from sitting-to-standing-to-sitting (from armchair) – no. (%) | | |
| Unable to perform function despite assistance from 2 people | | |
| Only able to perform function with assistance from 1 or 2 people | | |
| Able to perform function independently | | |
| Walking (with appropriate walking aid) – no. (%) | | |
| Unable to perform function despite assistance from 2 people | | |
| Only able to perform function with assistance from 1 or 2 people | | |
| Able to perform function independently | | |
| ≥ 4 metabolic equivalents | | |
| Co-existing disorders | | |
| Heart failure – no. (%) | | |
| NYHA score | | |
| 1 | | |
| 2 | | |
| 3 | | |
| 4 | | |
| Coronary artery disease – no. (%) | | |
| CCS score | | |
| Atrial flutter / fibrillation – no. (%) | | |
| Acute | | |
| Paroxysmal | | |
| Chronic | | |
| Diabetes – no. (%) | | |
| Dietary | | |
| Oral medication | | |
| Insulin | | |
| Obstructive sleep apnea – no. (%) | | |
| Apnea/Hypopnea Index (events / hour) | | |
| STOP BANG Score | | |
| Chronic obstructive pulmonary disease – no. (%) | | |
| Steroids use | | |
| Inhalation therapy | | |
| Use of noninvasive ventilation | | |
| Continuous positive airway pressure | | |
| Intensity of support (pressure level, cmH <sub>2</sub> O) | | |
| interiority of support (prosoure foreit, offit 120) | | |

#### eTable 2 – Additional Baseline Characteristics

| e l'able 2 – Additional Baseline Characteristics | | |
|---------------------------------------------------|-------------|------------|
| | Higher PEEP | Lower PEEP |
| Duration (hours / day) | (n = ) | (n = ) |
| Duration (hours / day) | | |
| Gastroesophageal reflux – no. (%) | | |
| ≥ 1 event/day | | |
| ≥ 1 event/week | | |
| ≥ 1 event/month | | |
| Respiratory infection within last month – no. (%) | | |
| Lower respiratory infection | | |
| Medications – no. (%) | | |
| Use of antibiotics (last 3 months) | | |
| Use of statins | | |
| Use of aspirin | | |
| Preoperative signs | | |
| FiO <sub>2</sub> , % | | |
| Temperature, °C | | |
| Tympanic – no. (%) | | |
| Nasal/oral – no. (%) | | |
| Bladder – no. (%) | | |
| Other | | |
| Preoperative laboratory tests | | |
| Blood gas obtained – no. (%) | | |
| Arterial – no. (%) | | |
| рН | | |
| PaO <sub>2</sub> , mmHg | | |
| PaCO <sub>2</sub> , mmHg | | |
| Hemoglobin, g/dL | | |
| INR | | |
| Creatinine, mg/dL | | |
| BUN, mg/dL | | |
| ALT, U | | |
| AST, U | | |
| Bilirubin, mg/dL | | |
| C-reactive protein, mg/L | | |
| Airway secretion – no. (%) | | |
| VAS dyspnea | | |
| VAS thoracic rest pain | | |
| VAS coughing pain | | |
| Spirometry obtained – no. (%) | | |
| Forced vital capacity, L | | |
| Predicted postoperative forced vital capacity, % | | |
| Forced expiratory volume at 1 second, L/1 sec | | |

#### eTable 2 - Additional Baseline Characteristics

| | Higher PEEP<br>(n = ) | Lower PEEP<br>(n = ) |
|---|---|---|
| Predicted postoperative forced expiratory volume at 1 second, % | | |
| Forced expiratory volume at 1 second / Forced vital capacity, % | | |
| Total lung capacity, L | | |
| Diffusing capacity for carbon monoxide | | |
| mmol/min/kPa | | |
| ml/min/mmHg | | |
| Predicted postoperative diffusing capacity for carbon monoxide, % | | |
| VO₂max (maximal oxygen consumption), mL/kg/min | | |
| Preoperative chest X-ray – no. (%) | | |
| Pulmonary infiltrates | | |
| Pleural effusion | | |
| Atelectasis | | |
| Pneumothorax | | |
| Cardiopulmonary edema | | |

Data are median (quartile 25th - quartile 75th) or N / total (%).

Abbreviations: PEEP is positive end-expiratory pressure; NYHA is New York Heart Association; INR is international normalized ratio; BUN is blood urea nitrogen; ALT is alanine transaminase; AST is aspartate transaminase; VAS is visual analogue scale.

Other

| eTable 3 – Additional Intraoperative | Characteristics | | | |
|---|---|---|---|---|
| · | Higher PEEP | Lower PEEP | Absolute Difference | p value |
| <u>-</u> | (n = ) | (n = ) | (95% CI) | p value |
| Patient position during induction – no. (%) | | | | |
| 0 – 15° | | | | |
| 15 - 30° | | | | |
| 30 - 45° | | | | |
| > 45° | | | | |
| Use of NIV for induction – no. (%) | | | | |
| Continuous positive airway pressure | | | | |
| NPPV | | | | |
| Method of one lung ventilation – no. (%) | | | | |
| Double lumen tube | | | | |
| Endobronchial blocker | | | | |
| Double lumen tube (embedded camera) | | | | |
| Other | | | | |
| Confirmation of OLV – no. (%) | | | | |
| Fiberoptic bronchoscopy | | | | |
| Embedded camera | | | | |
| Other | | | | |
| Patient positioning during surgery – no. (%) | | | | |
| Supine | | | | |
| Lateral | | | | |
| Prone | | | | |
| Other | | | | |
| Side of one lung ventilation – no. (%) | | | | |
| Left | | | | |
| Right | | | | |
| Side of surgery – no. (%) | | | | |
| Left | | | | |
| Right | | | | |
| Type of resection – no. (%) | | | | |
| Pneumectomy | | | | |
| Lobectomy | | | | |
| Wedge resection | | | | |
| Sleeve lobectomy | | | | |
| Segment resection | | | | |
| Pleurectomy | | | | |
| Other | | | | |
| Regional anesthesia | | | | |
| Epidural | | | | |
| Paravertebral | | | | |

#### eTable 3 - Additional Intraoperative Characteristics

| e rable 3 – Additional intraoperative | Onaracteristics | | | |
|---|---|---|---|---|
| | Higher PEEP | Lower PEEP | Absolute Difference | p value |
| <del>-</del> | (n = ) | (n = ) | (95% CI) | <u>, </u> |
| Neuromuscular monitoring – no. (%) | | | | |
| Surgical wound classification – no. (%) | | | | |
| Clean | | | | |
| Clean-contaminated | | | | |
| Contaminated | | | | |
| Dirty | | | | |
| Temperature at the end of the surgery, °C | | | | |
| Tympanic | | | | |
| Nasal/oral | | | | |
| Bladder | | | | |
| Other | | | | |
| Paralysis reversed | | | | |
| Residual curarization | | | | |
| Blood loss, mL | | | | |
| Urine output, mL | | | | |
| Continuation of ventilation – no. (%) | | | | |
| Reason | | | | |
| Hypothermia | | | | |
| Bleeding | | | | |
| Cardiovascular | | | | |
| Respiratory failure | | | | |
| Other | | | | |
| Duration, hours | | | | |
| Use of antibiotics – no. (%) | | | | |
| Prophylaxis | | | | |
| Th | | | | |

Data are median (quartile 25th - quartile 75th) or N / total (%).

Therapeutic

Abbreviations: PEEP is positive end-expiratory pressure; NIV is non-invasive ventilation; NPPV is non-invasive positive pressure ventilation; OLV is one lung ventilation.

Gelatine – no. (%)

| - | Higher PEEP | Lower PEEP | Absolute Difference | |
|---|---|---|---|---|
| | (n = ) | (n = ) | (95% CI) | p value |
| Analgesia | | | | |
| Alfentanyl – no. (%) | | | | |
| Dose, mg | | | | |
| Fentanyl – no. (%) | | | | |
| Dose, mg | | | | |
| Remifentanil – no. (%) | | | | |
| Dose, mg | | | | |
| Sufentanil – no. (%) | | | | |
| Dose, mg | | | | |
| Morphine – no. (%) | | | | |
| Dose, mg | | | | |
| Ketamine – no. (%) | | | | |
| Dose, mg | | | | |
| Volatiles | | | | |
| Desflurane – no. (%) | | | | |
| Dose, vol%*min | | | | |
| Sevoflurane – no. (%) | | | | |
| Dose, vol%*min | | | | |
| Sedatives | | | | |
| Dexmedetomidine – no. (%) | | | | |
| Dose, mg | | | | |
| Midazolam – no. (%) | | | | |
| Dose, mg | | | | |
| Propofol – no. (%) | | | | |
| Dose, mg | | | | |
| Thiopental – no. (%) | | | | |
| Dose, mg | | | | |
| Neuromuscular blocking agents | | | | |
| Atracurium – no. (%) | | | | |
| Dose, mg | | | | |
| Cisatracurium – no. (%) | | | | |
| Dose, mg | | | | |
| Rocuronium – no. (%) | | | | |
| Dose, mg | | | | |
| Succinylcholine – no. (%) | | | | |
| Dose, mg | | | | |
| Vecuronium – no. (%) | | | | |
| Dose, mg | | | | |
| Fluids | | | | |
| Hydroxyethyl starch – no. (%) | | | | |
| Dose, mL | | | | |

#### eTable 4 - Intraoperative Fluid and Drug Therapy

| | Higher PEEP (n = ) | Lower PEEP<br>(n = ) | Absolute Difference<br>(95% CI) | p value |
|---|---|---|---|---|
| Dose, mL | | (11 ) | (00 /0 01) | |
| Crystalloids – no. (%) | | | | |
| Dose, mL | | | | |
| Albumin – no. (%) | | | | |
| Dose, mL | | | | |
| Vasopressors | | | | |
| Ephedrine – no. (%) | | | | |
| Dose, mg | | | | |
| Adrenaline – no. (%) | | | | |
| Dose, mg | | | | |
| Noradrenaline – no. (%) | | | | |
| Dose, mg | | | | |
| Phenylephrine – no. (%) | | | | |
| Dose, mg | | | | |
| Blood products | | | | |
| Packed red blood cells - no. (%) | | | | |
| Dose, mL | | | | |
| Fresh frozen plasma – no. (%) | | | | |
| Dose, mL | | | | |
| Platelets – no. (%) | | | | |

Data are median (quartile 25th - quartile 75th) or N / total (%). Abbreviations: PEEP is positive end-expiratory pressure.

Dose, mL

#### PROTHOR Statistical Analysis Plan (v1.0, January 17th, 2024)

#### eTable 5 – Protocol Deviations

| | Higher PEEP<br>(n = ) | Lower PEEP<br>(n = ) | p value |
|---|---|---|---|
| Any protocol deviation – no. (%) | | | |
| SBP < 90mmHg unresponsive to fluids and/or vasoactive drugs | | | |
| New arrhythmias unresponsive to intervention (according to ACLS) | | | |
| Dosage of vasoactive drugs at the tolerance limit of the physician | | | |
| Need for massive transfusion | | | |
| Life-threatening surgical complication* | | | |
| Hypoxemia rescue** | | | |
| Hypercapnia rescue*** | | | |
| Deviation from prescribed PEEP | | | |
| Deviation from tidal volume | | | |
| Other | | | |

Data are median (quartile 25th - quartile 75th) or N / total (%).

 $\label{prop:permitting} \mbox{Abbreviations: PEEP is positive end-expiratory pressure.}$ 

<sup>\*</sup> Injury to the hemodynamic and respiratory system and brain, including major bleeding, tension pneumothorax, intracranial injury.

 $<sup>^{\</sup>star\star}$  Other than prescribed was necessary due to prolonged SpO2< 90%.

 $<sup>^{\</sup>star\star\star}$  Other than prescribed was necessary due to respiratory acidosis pH< 7.20

**Lower PEEP** 

(n = XXX)

**Absolute Difference** 

(95% CI)

p value

#### eTable 6 - Daily Assessment of Included Patients

| _ | Higher PEEP<br>(n = XXX) |
|-----------------------------------------|--------------------------|
| Day 1 | |
| Still in hospital – no. (%) | |
| Unplanned ICU admission – no. (%) | |
| New requirement of NIV or IMV – no. (%) | |
| New requirement of NIV – no. (%) | |
| Indication – no. (%) | |
| Standard of care | |
| Respiratory failure | |
| Other | |
| Type – no. (%) | |
| CPAP | |
| NPPV | |
| Other | |
| Pressure level, cmH <sub>2</sub> O | |
| Duration, hours | |
| New requirement of IMV – no. (%) | |
| Indication – no. (%) | |
| Resurgery | |
| Respiratory failure | |
| Other | |
| Duration, hours | |
| Physiotherapy – no. (%) | |
| Breathing exercises – no. (%) | |
| Incentive spirometry – no. (%) | |
| Cumulated ambulation score | |
| Day 2 | |
| Still in hospital – no. (%) | |
| Unplanned ICU admission – no. (%) | |
| New requirement of NIV or IMV – no. (%) | |
| New requirement of NIV – no. (%) | |
| Indication – no. (%) | |
| Standard of care | |
| Respiratory failure | |
| Other | |
| Type – no. (%) | |
| CPAP | |
| NPPV | |
| Other | |
| Pressure level, cmH <sub>2</sub> O | |
| Duration, hours | |
| New requirement of IMV – no. (%) | |
| Indication – no. (%) | |

Resurgery

p value

#### eTable 6 - Daily Assessment of Included Patients

CPAP

| e lable 6 – Dally Assessment of Inci | | | |
|---|---|---|---|
| | Higher PEEP<br>(n = XXX) | Lower PEEP<br>(n = XXX) | Absolute Difference<br>(95% CI) |
| Respiratory failure | | | |
| Other | | | |
| Duration, hours | | | |
| Physiotherapy – no. (%) | | | |
| Breathing exercises – no. (%) | | | |
| Incentive spirometry – no. (%) | | | |
| Cumulated ambulation score | | | |
| Day 3 | | | |
| Still in hospital – no. (%) | | | |
| Unplanned ICU admission – no. (%) | | | |
| New requirement of NIV or IMV – no. (%) | | | |
| New requirement of NIV – no. (%) | | | |
| Indication – no. (%) | | | |
| Standard of care | | | |
| Respiratory failure | | | |
| Other | | | |
| Type – no. (%) | | | |
| CPAP | | | |
| NPPV | | | |
| Other | | | |
| Pressure level, cmH2O | | | |
| Duration, hours | | | |
| New requirement of IMV – no. (%) | | | |
| Indication – no. (%) | | | |
| Resurgery | | | |
| Respiratory failure | | | |
| Other | | | |
| Duration, hours | | | |
| Physiotherapy – no. (%) | | | |
| Breathing exercises – no. (%) | | | |
| Incentive spirometry – no. (%) | | | |
| Cumulated ambulation score | | | |
| Day 4 | | | |
| Still in hospital – no. (%) | | | |
| Unplanned ICU admission – no. (%) | | | |
| New requirement of NIV or IMV – no. (%) | | | |
| New requirement of NIV – no. (%) | | | |
| Indication – no. (%) | | | |
| Standard of care | | | |
| Respiratory failure | | | |
| Other | | | |
| Type – no. (%) | | | |

#### eTable 6 - Daily Assessment of Included Patients

| | Higher PEEP<br>(n = XXX) | Lower PEEP<br>(n = XXX) | Absolute Difference<br>(95% CI) | p value |
|---|---|---|---|---|
| NPPV | , | , | , , | |
| Other | | | | |
| Pressure level, cmH <sub>2</sub> O | | | | |
| Duration, hours | | | | |
| New requirement of IMV – no. (%) | | | | |
| Indication – no. (%) | | | | |
| Resurgery | | | | |
| Respiratory failure | | | | |
| Other | | | | |
| Duration, hours | | | | |
| Physiotherapy – no. (%) | | | | |
| Breathing exercises – no. (%) | | | | |
| Incentive spirometry – no. (%) | | | | |
| Cumulated ambulation score | | | | |
| Day 5 | | | | |
| Still in hospital – no. (%) | | | | |
| Unplanned ICU admission - no. (%) | | | | |
| New requirement of NIV or IMV – no. (%) | | | | |
| New requirement of NIV – no. (%) | | | | |
| Indication – no. (%) | | | | |
| Standard of care | | | | |
| Respiratory failure | | | | |
| Other | | | | |
| Type – no. (%) | | | | |
| CPAP | | | | |
| NPPV | | | | |
| Other | | | | |
| Pressure level, cmH <sub>2</sub> O | | | | |
| Duration, hours | | | | |
| New requirement of IMV – no. (%) | | | | |
| Indication – no. (%) | | | | |
| Resurgery | | | | |
| Respiratory failure | | | | |
| Other | | | | |
| Duration, hours | | | | |
| Physiotherapy – no. (%) | | | | |
| Breathing exercises – no. (%) | | | | |
| Incentive spirometry – no. (%) | | | | |

Data are median (quartile 25th - quartile 75th) or N / total (%).

Cumulated ambulation score

Abbreviations: PEEP is positive end-expiratory pressure; ICU is intensive care unit; NIV is non-invasive ventilation; IMV is invasive mechanical ventilation; CPAP is continuous positive airway pressure; NPPV is non-invasive positive pressure ventilation

| eTable 7 - Additional Daily Assessn | nent of Included I | Patients | | |
|---|---|---|---|---|
| | Higher PEEP | Lower PEEP | Absolute Difference | n volue |
| _ | (n = XXX) | (n = XXX) | (95% CI) | p value |
| Day 1 | | | | |
| Impairment of wound healing – no. (%) | | | | |
| Superficial | | | | |
| Deep | | | | |
| Surgical wound infection – no. (%) | | | | |
| Superficial | | | | |
| Deep | | | | |
| Antibiotics – no. (%) | | | | |
| Therapeutically | | | | |
| PONV – no. (%) | | | | |
| Return of bowel function – no. (%) | | | | |
| Airway secretion – no. (%) | | | | |
| Purulent/yellow color | | | | |
| Not purulent | | | | |
| VAS dyspnea | | | | |
| VAS thoracic pain | | | | |
| VAS coughing pain | | | | |
| Day 2 | | | | |
| Impairment of wound healing – no. (%) | | | | |
| Superficial | | | | |
| Deep | | | | |
| Surgical wound infection – no. (%) | | | | |
| Superficial | | | | |
| Deep | | | | |
| Antibiotics – no. (%) | | | | |
| Therapeutically | | | | |
| PONV – no. (%) | | | | |
| Return of bowel function – no. (%) | | | | |
| Airway secretion – no. (%) | | | | |
| Purulent/yellow color | | | | |
| Not purulent | | | | |
| VAS dyspnea | | | | |
| VAS thoracic pain | | | | |
| VAS coughing pain | | | | |
| Day 3 | | | | |
| Impairment of wound healing – no. (%) Superficial | | | | |
| Deep | | | | |
| Surgical wound infection – no. (%) | | | | |
| Superficial | | | | |
| Deep | | | | |
| Antibiotics – no. (%) | | | | |
| Therapeutically | | | | |
| PONV – no. (%) | | | | |
| D (10. (70) | | | | |

Return of bowel function – no. (%)

#### eTable 7 - Additional Daily Assessment of Included Patients

| | Higher PEEP<br>(n = XXX) | Lower PEEP<br>(n = XXX) | Absolute Difference<br>(95% CI) | p value |
|---|---|---|---|---|
| Airway secretion – no. (%) | ( | ( | (************************************** | |
| Purulent/yellow color | | | | |
| Not purulent | | | | |
| VAS dyspnea | | | | |
| VAS thoracic pain | | | | |
| VAS coughing pain | | | | |
| Day 4 | | | | |
| Impairment of wound healing – no. (%) | | | | |
| Superficial | | | | |
| Deep | | | | |
| Surgical wound infection – no. (%) | | | | |
| Superficial | | | | |
| Deep | | | | |
| Antibiotics – no. (%) | | | | |
| Therapeutically | | | | |
| PONV – no. (%) | | | | |
| Return of bowel function – no. (%) | | | | |
| Airway secretion – no. (%) | | | | |
| Purulent/yellow color | | | | |
| Not purulent | | | | |
| VAS dyspnea | | | | |
| VAS thoracic pain | | | | |
| VAS coughing pain | | | | |
| Day 5 | | | | |
| Impairment of wound healing – no. (%) Superficial | | | | |
| Deep | | | | |
| Surgical wound infection – no. (%) | | | | |
| Superficial | | | | |
| Deep | | | | |
| Antibiotics – no. (%) | | | | |
| Therapeutically | | | | |
| PONV – no. (%) | | | | |
| Return of bowel function – no. (%) | | | | |
| Airway secretion – no. (%) | | | | |
| Purulent/yellow color | | | | |
| Not purulent | | | | |
| VAS dyspnea | | | | |
| VAS thoracic pain | | | | |
| VAS coughing pain | | | | |

Data are median (quartile 25th - quartile 75th) or N / total (%).

Abbreviations: PEEP is positive end-expiratory pressure; PONV is postoperative nausea and vomiting; VAS is visual analogue scale.

| e lable 8 – Dally Signs and Labo | d Laboratory of Included Patients | | | |
|---|---|---|---|---|
| | Higher PEEP<br>(n = XXX) | Lower PEEP<br>(n = XXX) | Absolute Difference<br>(95% CI) | p value |
| Day 1 | (11 7000) | (ii iii) | (0070 01) | |
| Respiratory rate, breaths/min | | | | |
| Heart rate, bpm | | | | |
| Mean arterial pressure, mmHg | | | | |
| Temperature, °C | | | | |
| Tympanic | | | | |
| Nasal/oral | | | | |
| Bladder | | | | |
| Other | | | | |
| SpO <sub>2</sub> , % | | | | |
| FiO <sub>2</sub> , % | | | | |
| Hemoglobin, g/dL | | | | |
| Creatinine, mg/dL Blood urea nitrogen, mg/dL | | | | |
| ALT, U | | | | |
| AST, U | | | | |
| Bilirubin, mg/dL | | | | |
| INR | | | | |
| C-reactive protein, g/L | | | | |
| Day 2 | | | | |
| Respiratory rate, breaths/min | | | | |
| Heart rate, bpm | | | | |
| Mean arterial pressure, mmHg | | | | |
| Temperature, °C | | | | |
| Tympanic | | | | |
| Nasal/oral | | | | |
| Bladder | | | | |
| Other | | | | |
| SpO <sub>2</sub> , % | | | | |
| FiO <sub>2</sub> , % | | | | |
| Hemoglobin, g/dL<br>Creatinine, mg/dL | | | | |
| Blood urea nitrogen, mg/dL | | | | |
| ALT, U | | | | |
| AST, U | | | | |
| Bilirubin, mg/dL | | | | |
| INR | | | | |
| C-reactive protein, g/L | | | | |
| Day 3 | | | | |
| Respiratory rate, breaths/min | | | | |
| Heart rate, bpm | | | | |
| Mean arterial pressure, mmHg | | | | |
| Temperature, °C | | | | |
| Tympanic | | | | |

Nasal/oral

| eTable 8 – Daily Signs and Laboratory of Included Patients | | | | |
|---|---|---|---|---|
| | Higher PEEP | Lower PEEP | Absolute Difference | n volue |
| | (n = XXX) | (n = XXX) | (95% CI) | <i>p</i> value |
| Bladder | | | | |
| Other | | | | |
| SpO <sub>2</sub> , % | | | | |
| FiO <sub>2</sub> , % | | | | |
| Hemoglobin, g/dL | | | | |
| Creatinine, mg/dL | | | | |
| Blood urea nitrogen, mg/dL | | | | |
| ALT, U | | | | |
| AST, U | | | | |
| Bilirubin, mg/dL | | | | |
| INR | | | | |
| C-reactive protein, g/L | | | | |
| Day 4 | | | | |
| Respiratory rate, breaths/min | | | | |
| Heart rate, bpm | | | | |
| Mean arterial pressure, mmHg | | | | |
| Temperature, °C | | | | |
| Tympanic | | | | |
| Nasal/oral | | | | |
| Bladder | | | | |
| Other | | | | |
| SpO <sub>2</sub> , % | | | | |
| FiO <sub>2</sub> , % | | | | |
| Hemoglobin, g/dL | | | | |
| Creatinine, mg/dL | | | | |
| Blood urea nitrogen, mg/dL | | | | |
| ALT, U | | | | |
| AST, U | | | | |
| Bilirubin, mg/dL | | | | |
| INR | | | | |
| C-reactive protein, g/L | | | | |
| Day 5 | | | | |
| Respiratory rate, breaths/min | | | | |
| Heart rate, bpm | | | | |
| Mean arterial pressure, mmHg | | | | |
| Temperature, °C | | | | |
| Tympanic | | | | |
| Nasal/oral | | | | |
| Bladder | | | | |
| Other | | | | |
| SpO <sub>2</sub> , % | | | | |
| FiO <sub>2</sub> , % | | | | |
| Hemoglobin, g/dL | | | | |
| Creatinine, mg/dL | | | | |

Blood urea nitrogen, mg/dL

#### PROTHOR Statistical Analysis Plan (v1.0, January 17th, 2024)

#### eTable 8 – Daily Signs and Laboratory of Included Patients

| | Higher PEEP<br>(n = XXX) | Lower PEEP<br>(n = XXX) | Absolute Difference<br>(95% CI) | p value |
|---|---|---|---|---|
| ALT, U | | | | |
| AST, U | | | | |
| Bilirubin, mg/dL | | | | |
| INR | | | | |
| C-reactive protein, g/L | | | | |

Data are median (quartile 25th - quartile 75th) or N / total (%).

Abbreviations: PEEP is positive end-expiratory pressure; INR is international normalized ratio; BUN is blood urea nitrogen; ALT is alanine transaminase; AST is aspartate transaminase.

#### eTable 9 - Day 1 Fluid and Drug Therapy

| erable 3 – Day 11 lala alla blug | | | | |
|---|---|---|---|---|
| | Higher PEEP | Lower PEEP | Absolute Difference | p value |
| | (n = ) | (n = ) | (95% CI) | p value |
| Fluids | | | | |
| Total fluid intake, mL | | | | |
| Hydroxyethyl starch – no. (%) | | | | |
| Dose, mL | | | | |
| Gelatin – no. (%) | | | | |
| Dose, mL | | | | |
| Crystalloids – no. (%) | | | | |
| Dose, mL | | | | |
| Albumin – no. (%) | | | | |
| Dose, mL | | | | |
| Vasopressors | | | | |
| Dobutamine – no. (%) | | | | |
| Dose, mg | | | | |
| Ephedrine – no. (%) | | | | |
| Dose, mg | | | | |
| Adrenaline – no. (%) | | | | |
| Dose, mg | | | | |
| Noradrenaline – no. (%) | | | | |
| Dose, mg | | | | |
| Phenylephrine – no. (%) | | | | |
| Dose, mg | | | | |
| Blood products | | | | |
| Packed red blood cells - no. (%) | | | | |
| Dose, mL | | | | |
| Fresh frozen plasma – no. (%) | | | | |
| Dose, mL | | | | |
| Platelets – no. (%) | | | | |

Data are median (quartile 25th - quartile 75th) or N / total (%). Abbreviations: PEEP is positive end-expiratory pressure.

Dose, mL

#### eTable 11 - Sensitivity Analyses for the Primary Outcome

| Higher PEEP | Lower PEEP | Odds Ratio | n valua |
|-------------|------------|------------|----------------|
| (n = XXX) | (n = XXX) | (95% CI) | <i>p</i> value |

Count events\*

Median (quartile 25th – quartile 75<sup>th</sup>)

Common effect GEE\*\*

Treatment-component interaction GEE\*\*\*

Average relative effect GEE\*\*\*\*

Abbreviations: CI is confidence interval; GEE is generalized estimating equations; PEEP is positive end expiratory pressure.

<sup>\* 95%</sup> confidence intervals calculated with proportional odds logistic regression and p values calculated Wilcoxon rank-sum test

<sup>\*\* 95%</sup> confidence intervals and p values calculated in a common effect GEE model (estimating a single treatment effect across all 10 components)

<sup>\*\*\*</sup> p value calculated in a GEE model (test whether the treatment effect differs across the 10 components)

<sup>\*\*\*\*</sup> p value calculated in a GEE model (estimating, then averaging, the 10 distinct treatment effects)

#### **PROPOSED FIGURE 1**

